CLINICAL TRIAL: NCT02725554
Title: Prospective, Randomized, Controlled, Multi-Center Study of Wireless Nerve Stimulation in the Treatment of Chronic Migraine
Brief Title: Study of Wireless Nerve Stimulation in the Treatment of Chronic Migraine
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was never initiated
Sponsor: Curonix LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30-00070
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Delayed Continuation Group (Active Comparator): All Subjects will be implanted with the StimRelieve HALO System. Subjects randomized to the delayed continuation group will have their systems deactivated until their 3 months follow-up visit. After this visit the stimulation will be reactivated.
  Interventions: Device: StimRelieve Halo System
- Continued Stim Group (Experimental): All Subjects will be implanted with the StimRelieve HALO System. Subjects randomized to the continued stim group will continue with active stimulation and monitored at defined intervals for data collection and device reprogramming, if needed.
  Interventions: Device: StimRelieve Halo System

INTERVENTIONS:
Device: StimRelieve Halo System — The StimRelieve Halo System is intended as the sole mitigating agent, or as an adjunct to other modes of therapy used in a multidisciplinary approach for chronic migraine as defined by the Third edition of the International Classification of headache disorders (ICDH-3). The system provides treatment by delivering small controlled electrical pulses to the occipital and supraorbital nerves, as it has been shown that for chronic migraine headaches the response to combined systems appears to be substantially better than occipital nerves stimulation alone.

SUMMARY:
The purpose of this study is to illustrate the safety and effectiveness of the StimRelieve Halo Nerve Stimulator System in the treatment of chronic migraine. The StimRelieve Halo System utilizes a minimally invasive procedure to implant a neurostimulator. This technology includes an octopolar electrode array stimulator with an embedded receiver. The energy source is a small, external, rechargeable transmitter, which is worn by the patient. The StimRelieve Halo System eliminates the implantable pulse generator, which has been the most common reason for reoperation or discomfort with existing devices.

For this study, all subjects will be randomized at enrollment into either a delayed or immediate continuation group. The immediate continuation group will immediately continue with the stimulation therapy after the 30-day trial period and will be monitored for a total of 12 months. The delayed activation group will have their device turned off after the 30-day trial period for the next 3-months. At the 3-month visit, both groups be evaluated and the delayed activation group will have their devices reactivated.

All subjects will immediately receive the permanent stimulator(s). The permanent stimulators can easily be removed if non-responders are identified. The wireless technology eliminates the need for externalized extensions, IPG's and thus reoperation. Additionally the outcome is highly dependent on placement of the stimulators. By eliminating the need for a staged trial, infection rates and incidence of pocket pain will decrease.

In this study, subjects will undergo a 30-day trial in order to demonstrate effectiveness. Immediate activation of all devices will be done in the post-op period based on sensory response and subject comfort. Subjects will be seen at 14-days post-implant to assess patient compliance with the device, assess clinical response and to adjust programming parameters if not responding. Subjects will be seen at 1 month post-implant and headache diaries and questionnaires will be reviewed. Subjects not responding to the therapy by at least a 30% reduction in headache days will be deemed non-responders and will be withdrawn from the study and can choose to have the device removed. After the trial period, all responders will follow their random assignment determined at enrollment (delayed or immediate continuation). All subjects will be monitored for a total of 13 months. Adverse events will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years but less than 65 years of age at time of informed consent;
* Subject who developed chronic migraine before the age of 60 years old;
* Subjects have been diagnosed with chronic migraine according to the International Classification of Headache Disorders-3 (ICHD-3) (2013) criteria;
* No medication overuse and not attributed to another causative disorder;
* Subjects have chronic migraine for at least 6 months prior to enrollment;
* Are refractory to conventional pharmacological chronic migraine treatments as defined by the failure to respond, or the intolerance, to at least 3 prophylaxis therapies (of which one is topiramate if not contraindicated) as determined by the investigator;
* Based on the medical opinion of the Principal Investigator, there is no evidence of anatomic abnormalities that could jeopardize the placement of the device or pose a hazard to the subject;
* Subject is willing to undergo surgical implant procedure, attend visits as scheduled, and comply with the study requirements;
* Based on the opinion of the Principal Investigator, subject is willing and able to operate the patient programmer, recharging equipment, and electronic diary equipment, and has the ability to undergo study assessments and provide accurate responses;
* Based on the opinion of the implanter, subject is a good surgical candidate for the implant procedure;
* Subject is male or non-pregnant female. If female of child-bearing potential, must have a negative pregnancy test at baseline visit, and if sexually active, must be using a medically acceptable method of contraception for the duration of their study participation; Subject is deemed to be neuropsychosocially appropriate for implantation therapies based of the assessment of a Clinical Psychologist, using face-to-face encounters and the psychological testing described in the measures.

Exclusion Criteria:

* Subject has undergone botulinum toxin (BOTOX) injections of the head and/or neck in the last 3 months;
* Subject is on prescribed opioid medication;
* Subject has a history of trigeminal autonomic cephalalgias;
* Subject has a history of other primary or secondary headache disorders;
* Subject has a history of trigeminal neuralgia;
* Subject has cranial postherpetic neuralgia (shingles);
* Subject has an active systemic infection or is immunocompromised; Insulin-dependent diabetic who is not controlled through diet and/or medication (determined by the physician) or non-insulin dependent diabetic who is not well controlled through diet and/or medication;
* Bleeding complications or coagulopathy issues;
* A life expectancy of less than one year;
* Any active implanted device whether turned off or on;
* Conditions requiring Magnetic Resonance Imaging (MRI) evaluation or diathermy procedures.
* Based on the medical opinion of the Principal Investigator, Psychologist and/or Psychiatrist, the subject has other psychological conditions (e.g., psychosis, suicidal ideation, borderline personality disorder, somatization, narcissism), other health conditions (e.g., substance abuse, another chronic condition requiring the regular use of opioid medication), or other legal concerns that would preclude his/her enrollment in the study or potentially confound the results of the study;
* Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device study while participating in this study;
* Subject is currently involved in litigation regarding injury, or is receiving worker's compensation benefits;
* Subject is currently being treated with repetitive transcranial magnetic stimulation r(TMS) or electro convulsion therapy (ECT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Headache Days | 3 Months
  The primary effectiveness endpoint is defined as a ≥ 30% reduction in headache days per month at 3 months post-trial with no increase in medication as compared to baseline.
Adverse Events | 12 Months
  The primary safety endpoint is the incidence and severity of adverse events through 3 months post-trial.

SECONDARY OUTCOMES:
Migraine Days | 3 Months
  Change in number of migraine days per month from baseline to 3 months post-trial
Headache Days | 3 Months
  Change in number of headache days per month from baseline to 3 months post-trial
Headache Impact Test (HIT) Score | 3 Months
  Change from baseline in total HIT-6 score to 3 months post-trial
Pain Medication | 3 Months
  Change from baseline in frequency of acute headache pain medication intake (all categories) at 3 months post-trial

IPD SHARING:
Plan to Share IPD: Yes
Within 6 months of end of study, data will be published. All study subject data will be anonymous.